CLINICAL TRIAL: NCT01030952
Title: A 3-week, Multi-center, Open-label, Randomized, Active-control, Parallel-group Study to Compare Effects of Nateglinide and Acarbose on Postprandial Glucose Fluctuation in Chinese Drug-naive Patients Type 2 Diabetes Mellitus
Brief Title: Effects of Nateglinide on Postprandial Glucose Excursion by Restoring Early Phase Insulin Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDJN608ACN07
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Nateglinide; Acarbose; glucose fluctuation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nateglinide; Acarbose

ARMS (2):
- Nateglinide (Experimental): Nateglinide tablets, oral administration, three times daily, 120 mg orally 10 minutes immediately before 3 meals three times daily.
  Interventions: Drug: Nateglinide
- Acarbose (Active Comparator): Acarbose tablets, oral administration, three times daily, dosage of 50 mg orally chewing with the first bite of a meal three times daily.
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Nateglinide — Nateglinide tablets, oral administration, three times daily, 120 mg orally 10 minutes immediately before 3 meals three times daily.
  Arms: Nateglinide
Drug: Acarbose — Acarbose tablets, oral administration, three times daily, dosage of 50 mg orally chewing with the first bite of a meal three times daily.
  Arms: Acarbose

SUMMARY:
A 3-week, multi-center, open-label, randomized, active-control, parallel-group study to compare effects of Nateglinide and Acarbose on postprandial glucose fluctuation in Chinese drug-naive patients type 2 diabetes mellitus (T2DM). In this study, participants in different groups took Nateglinide at a dose of 120 mg orally three times daily for up to 3 weeks or Acarbose at a dose of 50 mg three times daily for up to 3 weeks, respectively.

ELIGIBILITY:
Inclusion criteria

1. Patients must give written informed consent before any assessment is performed.
2. Male, non-fertile female or female of childbearing potential using a medically approved birth control method based on local regulations.
3. Drug naïve type 2 diabetes patients, defined as who neither take consecutive anti-hyperglycemic drug treatment more than 3 months anytime, nor any anti-hyperglycemic drug treatment in 4 weeks prior to visit 1.
4. Age in the range of 18-75 years inclusive.
5. HbA1c in the range of > 6.5 to ≤9.0% at Visit 1.

Exclusion criteria

1. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (>5 mIU/mL).
2. With known hypersensitivity to Nateglinide, Acarbose or any of the excipients.
3. A history of,

   1. type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, e.g., Cushing's syndrome and acromegaly.
   2. acute metabolic diabetic complications such as ketoacidosis or hyperosmolar state (coma) within the past 6 months.
   3. Torsades de pointes, sustained and clinically relevant ventricular tachycardia or ventricular fibrillation.
   4. percutaneous coronary intervention within the past 3 months.
   5. any of the following within the past 6 months: myocardial infarction (MI), coronary artery bypass surgery, unstable angina, or stroke.
4. Evidence of significant diabetic complications, e.g., symptomatic autonomic neuropathy or gastroparesis.
5. Acute infections which may affect blood glucose control within 4 weeks prior to visit 1.
6. Congestive heart failure requiring pharmacologic treatment. mg/dL (123μmol/L)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- China (3):
  - Sir Run Run Shaw Hospital, 3 East Qingchun Road, Hangzhou
  - Shanghai Tongji Hospital, 389 Xinchun Road, Shanghai
  - Shanghai Sixth People's Hospital, 600 Xuanshan Road, Shanghai

REFERENCES:
- [Background] Gao HW, Xie C, Wang HN, Lin YJ, Hong TP. Beneficial metabolic effects of nateglinide versus acarbose in patients with newly-diagnosed type 2 diabetes. Acta Pharmacol Sin. 2007 Apr;28(4):534-9. doi: 10.1111/j.1745-7254.2007.00534.x. PMID 17376293
- [Derived] Zhou J, Deng Z, Lu J, Li H, Zhang X, Peng Y, Mo Y, Bao Y, Jia W. Differential therapeutic effects of nateglinide and acarbose on fasting and postprandial lipid profiles: a randomized trial. Diabetes Technol Ther. 2015 Apr;17(4):229-34. doi: 10.1089/dia.2014.0299. PMID 25781235
- [Derived] Zhou J, Li H, Zhang X, Peng Y, Mo Y, Bao Y, Jia W. Nateglinide and acarbose are comparably effective reducers of postprandial glycemic excursions in chinese antihyperglycemic agent-naive subjects with type 2 diabetes. Diabetes Technol Ther. 2013 Jun;15(6):481-8. doi: 10.1089/dia.2013.0046. Epub 2013 Apr 30. PMID 23631607

RESULTS

PARTICIPANT FLOW:
Groups:
- Nateglinide: 120 mg by mouth, three times daily 10 minutes immediately before 3 meals
- Acarbose: patients in Acarbose group received Acarbose 50 mg by mouth, three times daily with the first bite of a meal
Period: Overall Study
Arm/Group | Nateglinide | Acarbose
Started | 51 | 52
Completed | 49 | 49
Not Completed | 2 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Informed consent withdrawal | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Unexplained | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nateglinide | Acarbose | Total
Number analyzed (Participants) | 51 | 52 | 103
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.34) | 53.7 (9.36) | 53.5 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 (39.22) | 23 (44.23) | 43
  Male | 31 (60.78) | 29 (55.7) | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Area Under Curve of 0-4 Hours Postprandial Glucose (AUCpp0-4hours) in Standardized Meal Test Using Continuous Glucose Monitoring System (CGMS)
Description: The postprandial glucose area under the curve (AUC)was calculated using values from the 3 time points. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM.
  0-4 hours AUC were calculated using trapezoid methods.
Time Frame: 3 weeks (end of study) minus baseline
Population: Intent to Treat population - All patients who received at least one dose of study drug after random allocation and had at least one primary or secondary efficacy evaluation after baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimoles hours per litre (mmol*hr/L)
Groups:
- Nateglinide: 120 mg by mouth, three times daily (P.O. t.i.d) 10 minutes immediately before 3 meals
- Acarbose: 50 mg by mouth, three times daily (P.O. t.i.d) with the first bite of a meal
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 39 | 42
millimoles hours per litre (mmol*hr/L) | -9.20 (11.71) [-11.780 to -6.621] | -9.92 (9.97) [-12.407 to -7.438]

2. Secondary Outcome: Change in Incremental Glucose Peak (IGP) From Baseline
Description: Incremental glucose peak (IGP) was the maximal incremental increase in blood glucose obtained at any point after meal
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/L)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
millimoles per litre (mmol/L) | -2.72 (2.86) | -1.89 (2.76)

3. Secondary Outcome: Change in Mean Blood Glucose (MBG)
Description: The 24 hour mean blood glucose (MBG) level was calculated as the mean of all the consecutive readings on baseline and end of study(3 weeks later) separately.
Time Frame: baseline and at 3 weeks (end of study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/l)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
millimoles per litre (mmol/l) | -1.16 (1.24) | -0.78 (1.29)

4. Secondary Outcome: Change in Standard Deviation (SD) From Baseline of Mean Blood Glucose (MBG) Over 24 Hours.
Description: Change in standard deviation (SD) from baseline of mean blood glucose (MBG) describes the range of blood glucose fluctuation over 24 hours.
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
mmol/l | -0.48 (0.63) | -0.63 (0.59)

5. Secondary Outcome: Change in Mean of Daily Difference of Paired Blood Glucose Value (MODD)
Description: The mean of the daily differences (MODD), calculated as the average absolute difference of paired glucose values during two successive 24 hour periods, was used to assess day-to-day glycaemic variability.
Time Frame: baseline, 3 weeks (end of study)
Population: Intent-to treat population (ITT): All randomized participants who received at least 1 dose of study drug, had valid baseline data, and at least 1 post-baseline assessment of the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/l)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
millimoles per litre (mmol/l) | -0.06 (0.95) | -0.21 (0.86)

6. Secondary Outcome: Changes in 24 Hour Glucose Area Under Curve (AUCpp)
Description: Blood samples were collected for measurement of plasma glucose at 30, 60, 90, and 120 minutes following the start of a standardized meal test at Baseline and Week 4. The postprandial glucose area under the curve was calculated using values from the 4 time points. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM.
Time Frame: baseline, end of study (3 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol*min/L
Groups:
- Nateglinide: 120 mg by mouth, three times daily (P.O. t.i.d.) 10 minutes immediately before 3 meals
- Acarbose: 50 mg by mouth, three times daily (P.O. t.i.d.) with the first bite of a meal
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
mmol*min/L | -1.16 (1.24) | -0.78 (1.29)

7. Secondary Outcome: Change in Glycated Serum Albumin (GSA) Levels From Baseline After Treatment
Description: GSA levels were to be determined by CGMS at 7:00~10:00 am in the 4-hour standardized meal test before treatment after overnight fasting for efficacy assessments
Time Frame: baseline, 3 weeks (end of study)
Population: Intent to Treat population - All patients who received at least one dose of study drug after random allocation and had at least one primary or secondary efficacy evaluation after baseline. During different time points, participants with observations at that time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 51
percent | -2.22 (1.90) | -1.74 (1.50)

8. Secondary Outcome: Change in Insulin Levels (μU/ml) During Standardized Meal Test at Endpoint From Baseline
Description: This outcome measure calculated the change in insulin levels between groups over time at 0, 30 then 120 minutes
Time Frame: baseline, 3 weeks (end of study)
Population: The Intent to Treat (ITT) population consists of all patients randomized and who have at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: (μU/ml)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
(μU/ml)
  0 minutes | 0.32 (5.88) | -0.21 (3.16)
  30 minutes | 13.87 (20.98) | -6.64 (6.44)
  120 minutes | 15.03 (31.22) | -16.24 (22.01)

9. Secondary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: change in LDL-C at 0, 30 and 120 minutes
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/l)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
millimoles per litre (mmol/l)
  0 minutes | -0.04 (0.65) | 0.064 (0.44)
  30 minutes | -0.06 (0.63) | 0.09 (0.44)
  120 minutes | -0.04 (0.56) | 0.13 (0.42)

10. Secondary Outcome: Change of Total Cholesterol in Blood Lipids Levels During Standardized Meal Test at Endpoint From Baseline at Each Time Point
Description: time to change in Total Cholesterol blood lipids level at 0, 30, 120 minutes
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/l)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
millimoles per litre (mmol/l)
  0 minutes | -0.03 (0.67) | -0.09 (0.55)
  30 minutes | -0.06 (0.70) | 0.56 (0.04)
  120 minutes | -0.01 (0.61) | 0.03 (0.68)

11. Secondary Outcome: Change in Triglyceride (TG)Levels in Blood Lipid Levels During Standardized Meal Test at Endpoint
Description: TG change in blood lipids level from baseline to endpoint
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/l)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
millimoles per litre (mmol/l)
  0 minutes | -0.19 (0.63) | -0.48 (1.16)
  30 minutes | -0.23 (0.68) | -0.39 (0.81)
  120 minutes | -0.19 (0.83) | -0.47 (1.02)

12. Secondary Outcome: Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) at the End of the Study
Description: Blood samples were collected for measurement of HDL-C prior to (fasting) and 120 minutes following the start of a standardized meal test at Baseline and Week 3. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. HDL-C was assessed at each study site using the same method and same reference value.
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/l)
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
millimoles per litre (mmol/l)
  0 minutes | 0.20 (0.10) | -0.02 (0.31)
  30 minutes | 0.02 (0.10) | 0.01 (0.16)
  120 minutes | 0.03 (0.09) | 0.00 (0.17)

13. Secondary Outcome: Change in Mean Amplitude of Glycaemic Excursion (MAGE)
Description: mean amplitude of glycaemic excursion (MAGE) is an average of the amplitudes of all glycemic excursions greater than a prespecified threshold size
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 51 | 52
mmol/l | 5.27 (2.09) | 5.03 (1.82)

14. Secondary Outcome: The Percent of 24 Hour Hypoglycemic Measurements
Description: Measures/compares changes in percentage of hypoglycemia(<3.9mmol/l or <70 mg/dl) in glucose measurements in 24hours by continuous glucose monitoring system (CGMS) at endpoint from baseline between groups. Reported values are percent change of the base absolute values [100% * ((X-Y)/Y)]
Time Frame: baseline, 3 weeks (end of study)
Population: Intent-to-treat population (ITT): All randomized participants who received at least 1 dose of study drug, had valid baseline data, and at least 1 post-baseline assessment of the primary efficacy variable. During different time points, participants with observations at that time point were included in the analysis
Measure: Mean (Standard Deviation); unit: percent of measurements
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 39 | 42
percent of measurements | 0.82 (2.22) | -0.57 (1.77)

15. Secondary Outcome: Change in Percent of 24 Hour Hyperglycemic Measurements
Description: Measures/compares changes in percentage of hyperglycemia (>7.8mmol/l or 140 mg/dl) in glucose measurements in 24 hours by continuous glucose monitoring system (CGMS) at endpoint from baseline between groups. Reported values are percent change of the base absolute values [100% * ((X-Y)/Y)]
Time Frame: baseline, 3 weeks (end of study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of measurements
Arm/Group | Nateglinide | Acarbose
Number analyzed (Participants) | 39 | 42
percent of measurements | -50.83 (64.62) | -33.82 (75.39)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Nateglinide | Acarbose
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 7/51 | 16/52
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nateglinide (N=51) | Acarbose (N=52)
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Frequency bowel movements (Gastrointestinal disorders) | 0 | 2
Gastrointestinal flatulence (Gastrointestinal disorders) | 0 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
White blood cells count decrease (Investigations) | 0 | 1
White blood cells count increase (Investigations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
White blood cells urine positive (Investigations) | 0 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.